CLINICAL TRIAL: NCT06190613
Title: Adapting and Testing a Combination Peer Navigation and MHealth Intervention to Enhance Treatment Engagement and Viral Suppression Among Sexual and Gender Minority Youth in Nigeria
Brief Title: Combination Intervention to Enhance Treatment Engagement and Viral Suppression Among Sexual and Gender Minority Youth in Nigeria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Kuhns, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: iCARE R34; 1R34MH132453 (NIH)
Record Dates: First submitted 2023-12-13; First posted 2024-01-05 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination peer navigation and mHealth Intervention (Other): Peer navigation and SMS text message medication reminders
  Interventions: Behavioral: Combination Peer navigation and mHealth intervention
- Control (No Intervention): standard of care

INTERVENTIONS:
Behavioral: Combination Peer navigation and mHealth intervention — Peer navigation and SMS text message medication reminders (adapted to YMSM and YTW in community outreach-based delivery approach)
  Arms: Combination peer navigation and mHealth Intervention

SUMMARY:
The study will adapt and test a combination peer navigation and mHealth approach, Intensive Combination Approach to Rollback the Epidemic in Nigeria (iCARE Nigeria), to improve HIV treatment engagement, medication adherence and viral suppression among YMSM and YTW, ages 15-29.

DETAILED DESCRIPTION:
The study will adapt and test a combination peer navigation and mHealth approach, Intensive Combination Approach to Rollback the Epidemic in Nigeria (iCARE Nigeria), to improve HIV treatment engagement, medication adherence and viral suppression among young men who have sex with men (YMSM) and young transgender women (YTW), ages 15-29. The 24-week pilot study will randomize participants at a ratio of 1:1 to the intervention or control. The goals of the pilot study are to assess: a) whether the intervention worked as intended (initial efficacy); and b) the feasibility, satisfaction, and acceptability among the target population of YMSM and YTW receiving HIV care in the community setting.

Specific aims are to:

1. Adapt the iCARE Nigeria HIV clinic-based intervention to a community-based outreach approach for YMSM and YTW ages 15-29 in Ibadan, Nigeria. This process will be structured using best practices for adaptation of evidence-based intervention, including distillation of adaptable components and incorporation of feedback from stakeholders, following user-centered principles of iterative design.
2. In a randomized controlled trial, test the adapted iCARE intervention for initial efficacy, feasibility, satisfaction, and acceptability among YMSM and YTW in the key population (KP)-focused community settings. The primary outcome will be viral load suppression (viral load<200 copies/mL). Secondary outcomes include antiretroviral drug adherence, and treatment retention via abstraction of medical records.
3. Evaluate implementation indicators based on RE-AIM (reach, adoption, implementation, maintenance) to improve external validity and to inform sustainability and scalability of the adapted iCARE Nigeria intervention. A mixed methods approach will be used to collect data for implementation outcomes from interventionists, intervention participants, and representatives of KP-friendly community centers.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* registered as a patient at one of the collaborating key population (KP)-focused community centers
* male sex at birth
* identify as YMSM or YTW (or report a history of sex with men)
* on ART for at least 3 months
* understand and read basic English, Yoruba, or Pidgin English
* intention to remain a patient at a collaborating clinic during the 24-week follow-up period
* has a cellphone

Exclusion Criteria:

* Unable to obtain parental permission if 15 years of age and not emancipated

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — identify as YMSM or YTW
Enrollment: 100 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
HIV viral load suppression | Baseline, 24 weeks
  Viral load suppression (<200 copies/mL) at baseline and 24 weeks

SECONDARY OUTCOMES:
Retention in HIV care | Baseline, 24 weeks
  Two medical visits in the 24-week study period, with a minimum of 60 days between visits
Medication adherence | Baseline, 24 weeks
  Self-reported measure of adherence on visual analogue scale (0-100), with adherence measured as >or = 90%
Feasibility of intervention | 24 weeks
  Phone-related and SMS text-related problems resulting in <10% message failure, measured by text message platform administrative reports
Acceptability of intervention | 24 weeks
  Acceptability report of >90% agreement based on Client Satisfaction Questionnaire-8 (CSQ-8)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Kuhns, PhD, Principal Investigator — Northwestern University
Locations (1):
- University of Ibadan, Ibadan, Nigeria

IPD SHARING:
Plan to Share IPD: No